CLINICAL TRIAL: NCT05020132
Title: Prospective Evaluation of Bowel Dysfunction After Rectal Cancer Treatment
Brief Title: Bowel Dysfunction After Rectal Cancer Treatment
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Hospital Universitari MútuaTerrassa (Unknown)
Responsible Party: Principal Investigator, Yolanda Ribas, Principal Investigator, Consorci Sanitari de Terrassa
Other Study IDs: LARS
Record Dates: First submitted 2021-08-17; First posted 2021-08-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bowel dysfunction after rectal cancer treatment may significantly affect the quality of life. Our study aimed to estimate the incidence and characterize the Low Anterior Resection Syndrome(LARS). We performed a prospective evaluation of patients treated with anterior resection for rectal cancer at two hospitals. Assessment was performed at baseline, after neoadjuvant treatment, and 1, 6 and 12 months after bowel transit reconstruction using the following scores: Bristol scale, LARS score, MSK-BFI, FIQL, EORTC-QLQ30 and a visual analogue scale.

DETAILED DESCRIPTION:
Low anterior resection syndrome (LARS) refers to wide-ranging symptoms including evacuatory dysfunction, fecal urgency and incontinence. The assessment of bowel dysfunction after rectal cancer treatment has improved since the development of the LARS score. This score has widely been used with a meta-analysis reporting a pooled prevalence of "major LARS" of 41%. However, several studies have found a large proportion of patients with major LARS in the general population without rectal cancer raising questions about the specificity of this score. Moreover, most studies on the prevalence of LARS do not include a baseline evaluation and, therefore, may not allow establishing whether the dysfunctions appeared after the treatment. Consequently, we considered that a prospective study including a baseline evaluation and multiple validated questionnaires was required. The present study aimed to estimate the incidence and characterize bowel dysfunction after rectal cancer treatment. The results of this study will be useful to improve the preoperative information given to the patient and the shared decision-making process.

ELIGIBILITY:
Inclusion Criteria:

Patients with anterior resection for rectal adenocarcinoma with curative intention, with or without neoadjuvant chemoradiotherapy, total or partial excision of the mesorectum, colorectal or coloanal anastomosis.

Exclusion Criteria:

* disseminated disease
* surgery with palliative intent
* refusal to participate in the study
* intellectual difficulty to answer the questionnaires

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anterior resection for rectal adenocarcinoma with curative intention, with or without neoadjuvant chemoradiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in the LARS score between baseline and 12 months | 12 months
  Change in the LARS score (Low Anterior Resection Score) between baseline and 12 months after bowel transit reconstruction (primary surgery or ileostomy closure). The LARS score is a 5-item scoring system which classifies patients into three severity categories: no LARS (0-20 points), minor LARS (21-29 points), and major LARS (30-42 points). A higher score represents worse bowel function. This score also includes a question about the impact on quality of life.
Change in the MSK-BFI between baseline and 12 months (MSK-BFI) | 12 months
  Change in the Memorial Sloan-Kettering Cancer Center Bowel Function Instrument (MSK-BFI) between baseline and 12 months after bowel transit reconstruction (primary surgery or ileostomy closure). The MSK-BFI includes 18 questions with five frequency options ranging from never through to always. A total score and three subscales (frequency, diet, and urgency) can be calculated. A higher score represents better bowel function.
Change in the Bristol stool chart between baseline and 12 months | 12 months
  Change in the Bristol stool chart between baseline and 12 months after bowel transit reconstruction (primary surgery or ileostomy closure). The Bristol stool chart shows seven categories of stool. The Bristol score was subclassified into three categories: Bristol 1-2 (hard stools), Bristol 3-4 (normal stools), and Bristol 5-7 (loose or liquid stools).

SECONDARY OUTCOMES:
Change in the Visual Analogue Scale (VAS) between baseline and 12 months | 12 months
  Change in the Visual Analogue Scale (VAS) between baseline and 12 months after bowel transit reconstruction (primary surgery or ileostomy closure). The VAS ranges from 0 (worst bowel function) to 10 (best)
Change in the EORTC QLQ-C30 between baseline and 12 months | 12 months
  Change in the European Organization for Research and Treatment of Cancer Quality oF Life Questionnaire (EORTC QLQ-C30) between baseline and 12 months after bowel transit reconstruction (primary surgery or ileostomy closure). The EORTC QLQ-C30 is a self-administered questionnaire developed to assess the quality of life of patients with cancer. The global QoL scale and 5 functional scales (physical, role, cognitive, emotional, and social functioning) can be calculated. All scales range from 0 to 100. A higher score for the global health status represents a higher quality of life, and a higher score for a functional scale represents a higher / healthy level of functioning.
Change in the Fecal Incontinence Quality of Life (FIQL) between baseline and 12 months | 12 months
  Change in the Fecal Incontinence Quality of Life (FIQL) between baseline and 12 months after bowel transit reconstruction (primary surgery or ileostomy closure). The FIQL score includes 29 items which form four scales: lifestyle, coping/behavior, depression/self-perception, and embarrassment. Scores range from 0 to 4 and a higher value represents a better quality of life.
Correlation of the severity of LARS with the quality of life | 12 months
  Correlation of the severity of LARS (LARS score and MSK-BFI) with the quality of life (EORTC QLQ-C30)
Multivariate analysis of risk factors for LARS | 12 months
  Assessment of independent predictors of the LARS score at the 12-month visit in a multiple linear regression model. Univariate linear regression analysis was initially performed to identify the demographic, clinical and surgical factors associated with the 12-month LARS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari de Terrassa, Terrassa, Barcelona, Spain